CLINICAL TRIAL: NCT02706548
Title: Feasibility of the Integrative Medication Self-Management Intervention to Promote Medication Adherence
Acronym: IMedS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Milwaukee (Other)
Responsible Party: Principal Investigator, Jaclyn Schwartz, Doctoral Student, University of Wisconsin, Milwaukee
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15.048
Record Dates: First submitted 2016-03-08; First posted 2016-03-11 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Medication Adherence; Chronic Disease
Keywords: occupational therapy; medication adherence; intervention studies
MeSH Terms: conditions — Medication Adherence; Chronic Disease | interventions — Methods

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Occupational Therapy Intervention Group (Experimental): Thirty-minute intervention in which the participant and interventionist discuss past medication taking performance, medication-related goals, and strategies to meet goals. Intervention is enhanced with motivational interviewing and therapeutic use of self.
  Interventions: Behavioral: Integrative Medication Self Management (IMedS) Intervention
- Standard Care Intervention Group (Active Comparator): Thirty-minute educational intervention in which the participant and interventionist review a pamphlet on adherence to medication.
  Interventions: Behavioral: Standard Care Educational Intervention

INTERVENTIONS:
Behavioral: Integrative Medication Self Management (IMedS) Intervention — Half of participants received a manualized 30-minute occupational therapy intervention, Integrative Medication Self-Management Intervention (IMedS). During IMedS, the interventionist and client progress through three steps in which the pair: 1) reflect on past performance of medication management, 2) set a medication goal, and 3) generate strategies to reach the goal. During strategy generation, the interventionist uses therapeutic use of self and motivational interviewing to help the client self-generate new medication management strategies, specifically addressing 1) altering the activity, 2) advocacy, 3) education, 4) assistive technology, 5) environmental modifications, and 6) securing timely refills.
  Arms: Occupational Therapy Intervention Group
Behavioral: Standard Care Educational Intervention — The standard care educational intervention was a 30-minute pamphlet based educational session. In the standard care intervention group, participants and interventionist first reviewed the pamphlet, Managing Your Medicines: Our Guide to Effective Medication Management (American Heart Association & American Stroke Association, 2013). Then, the interventionist engaged in active listening, where she asked open-ended questions about the participant's medication routines and provided simple reflections. For the standard care procedures, the interventionist was prohibited from providing affirmations, complex reflections, summaries, problem-solving, or suggesting any specific interventions.
  Arms: Standard Care Intervention Group

SUMMARY:
Many persons with chronic health conditions fail to take their medications as prescribed, resulting in declines in health and function. Unfortunately, current interventions for medication nonadherence are not very effective. This objective of this study is to test a new intervention, the Integrative Medication Self-management (IMedS) intervention to improve medication adherence in adults with chronic health conditions.

DETAILED DESCRIPTION:
Many persons with chronic health conditions fail to take their medications as prescribed, resulting in declines in health and function. Objective: The purpose of this study was to perform a phase I feasibility study to understand if an integrated occupational therapy intervention could help people with chronic health conditions improve their adherence to medications. Method: Using a small-N design, we report single-subject analyses of the medication adherence, behavior counts, and perceptions of medication adherence of participants before and after either an occupational therapy intervention or standard of care intervention. We used a multiple baseline approach with inter-subject replication, and blinding.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with a chronic health condition
* Live in the community
* A medication regimen of 5 or more medications a day recommended by a health care professional
* Independently manage medications
* Difficulty taking medications as prescribed
* Live in the Milwaukee area

Exclusion Criteria:

* Significant cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-10; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Medication Adherence | 4 Weeks
  Daily medication possession ratio via diary
Self-perceived improvements in ability to mange medications | 4 weeks
  Participants at the end of the study indicate if they believe that their ability to manage medications has improved, declined, or stayed the same.

SECONDARY OUTCOMES:
Strategies used to manage medications | 4 weeks
  Number of new strategies in daily life used to manage medications per participant report

IPD SHARING:
Plan to Share IPD: Yes
Single-subject data available in publications

REFERENCES:
- [Result] Schwartz JK, Smith RO. Benefits of Student Engagement in Intervention Research. Am J Occup Ther. 2015 Sep-Oct;69 Suppl 2:6912185050p1-6912185050p10. doi: 10.5014/ajot.2015.018200. PMID 26539678
- [Derived] Schwartz JK, Smith RO. Intervention Promoting Medication Adherence: A Randomized, Phase I, Small-N Study. Am J Occup Ther. 2016 Nov/Dec;70(6):7006240010p1-7006240010p11. doi: 10.5014/ajot.2016.021006. PMID 27767947